CLINICAL TRIAL: NCT00321867
Title: Porcine-Derived Small Intestine Submucosa Graft-Augmented Rectocele Repair-A Randomized Trial
Brief Title: Graft-Augmented Rectocele Repair-A Randomized Surgical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Vivian Sung, Principal Investigator, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-0086
Record Dates: First submitted 2006-05-03; First posted 2006-05-04 (Estimated); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Rectocele
Keywords: rectocele; pelvic prolapse; graft; surgical repair
MeSH Terms: conditions — Rectocele

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Native tissue repair
  Interventions: Procedure: Control
- 2 (Experimental): Posterior repair with graft
  Interventions: Procedure: Graft augmented posterior repair

INTERVENTIONS:
Procedure: Graft augmented posterior repair — Posterior repair with graft
  Arms: 2
Procedure: Control — Native tissue repair
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether adding a graft during a rectocele repair will improve the success rate of the repair.

DETAILED DESCRIPTION:
Rectoceles may have a significant effect on the quality of life of women. Symptoms associated with rectoceles include a protruding vaginal mass, persistent pelvic pressure, and sexual dysfunction. Surgical repair is the most common treatment with success rates ranging from 65%-85% at 1-2 years. In an attempt to improve surgical outcomes, clinicians are using graft materials to augment weakened tissues in rectocele repairs: however, there is little data to support or refute these practices. The purpose of this study is to estimate the effect of graft augmentation on objective and subjective outcomes.

Comparison: Rectocele repair without graft, compared to rectocele repair with the SurgiSIS (TM) graft.

ELIGIBILITY:
Inclusion Criteria:

* Women with stage 2 or greater symptomatic rectocele
* Women electing to undergo surgical rectocele repair
* Women over age 21 years
* Women willing to comply with study procedures and follow-up

Exclusion Criteria:

* Pregnant or nursing women
* History of porcine allergy
* History of connective tissue disease, pelvic malignancy, or pelvic radiation
* Women undergoing concurrent sacral colpopexy

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2004-01; Primary Completion 2010-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Anatomic cure defined by standardized POPQ measures | 12 months

SECONDARY OUTCOMES:
Quality of life based on PFIQ validated questionnaire | 12 months
Sexual function | 12 months
Patient centered goals | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vivian W Sung, MD MPH, Principal Investigator — Women and Infants Hospital
Locations (1):
- Women and Infants Hospital of Rhode Island, Providence, Rhode Island, United States

REFERENCES:
- [Result] Sung VW, Rardin CR, Raker CA, Lasala CA, Myers DL. Porcine subintestinal submucosal graft augmentation for rectocele repair: a randomized controlled trial. Obstet Gynecol. 2012 Jan;119(1):125-33. doi: 10.1097/AOG.0b013e31823d407e. PMID 22183220
- [Derived] Yeung E, Baessler K, Christmann-Schmid C, Haya N, Chen Z, Wallace SA, Mowat A, Maher C. Transvaginal mesh or grafts or native tissue repair for vaginal prolapse. Cochrane Database Syst Rev. 2024 Mar 13;3(3):CD012079. doi: 10.1002/14651858.CD012079.pub2. PMID 38477494